CLINICAL TRIAL: NCT06388395
Title: Clinical Performance of Mandibular All-on-4 Modified Polyetheretherketone Treatment Approach Versus Conventional Metal Framework and Hybrid Prostheses: a Randomized Clinical Trial
Brief Title: Clinical Performance of All-on-4 PEEK and Conventional Prostheses
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ahmed Aziz, Assistant Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-23-05-12-02-F
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Failure, Prosthesis; Dental Prosthesis, Implant-Supported; Survival, Prosthesis; Complete Edentulism; Complication;Prostheses
MeSH Terms: conditions — Prosthesis Failure | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Two groups will be provided with two types of implant-supported prostheses
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Block randomization will be used to randomly assign participants. The sequences will be concealed in opaque, consecutively numbered envelopes for each block. One envelope will be obtained for each participant, corresponding to the assignment of the protocol (conventional versus PEEK). The outcome assessor will be independent and not involved in any treatment procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Accuracy of full-arch surgical guides (Experimental): Two surgical guides (milled and 3D printed) will be used randomly to assess the accuracy of the guides following guided implant surgery.
  Interventions: Procedure: Accuracy of full-arch surgical guides
- Survival and complications of the prostheses (Experimental): The clinical performance of the two different treatment concepts during the follow up period of 3 years concerning screw loosening, veneering material chipping, wear or staining, prosthesis survival and success will be assessed.
  Interventions: Procedure: Survival and complications of the prostheses
- Survival and complications of the implants (Experimental): The implants survival and success rates will be evaluated after 1, 2 and 3 years of prostheses insertion.
  Interventions: Procedure: Survival and complications of the implants
- Conventional implant-supported prosthesis (Experimental): Full-arch implant-supported conventional (metal-resin) prosthesis will be constructed and assessed for up to 3 years
  Interventions: Procedure: Conventional (metal-resin) implant-supported prosthesis
- PEEK implant-supported prosthesis (Experimental): Full-arch implant-supported PEEK prosthesis will be constructed and assessed for up to 3 years
  Interventions: Procedure: PEEK implant-supported prosthesis

INTERVENTIONS:
Procedure: Accuracy of full-arch surgical guides — The accuracy of the surgical guides will be assessed by superimposing the pre and post-treatment CBCT scans.
  Arms: Accuracy of full-arch surgical guides
Procedure: Survival and complications of the prostheses — Two different prostheses will be assessed (conventional and PEEK). All complications will be recorded for a period of 3 years
  Arms: Survival and complications of the prostheses
Procedure: Survival and complications of the implants — The effect of the two different prostheses on implants will be assessed in terms of survival and success rates.
  Arms: Survival and complications of the implants
Procedure: Conventional (metal-resin) implant-supported prosthesis — Full-mouth implant-supported conventional prosthesis will be constructed and evaluated for up to 3 years.
  Arms: Conventional implant-supported prosthesis
Procedure: PEEK implant-supported prosthesis — Full-mouth implant-supported PEEK prosthesis will be constructed and evaluated for up to 3 years.
  Arms: PEEK implant-supported prosthesis

SUMMARY:
The all-on-4 treatment approach for completely edentulous mandible is a proven concept. However, there are still issues regarding the use of metal substructure to support the prostheses such as allergy, metallic taste, and aesthetic. Therefore, other materials such as polyetheretherketone (PEEK) are being tested for its suitability and is showing good potential. However, available evidence is limited regarding its clinical performance. Thus, the aim of this study is to compare clinical performance of all-on-4 treatment concept utilizing PEEK versus conventional metal framework as substructure in fully edentulous mandible. Thirty suitable patients will receive either PEEK or conventional all-on-4 prostheses for fully edentulous mandible. The prostheses will be retained by four implants utilizing the all-on-4 principle. Clinical performance will be assessed during the follow up period of up 3 years concerning screw loosening, material chipping or fracture, wear or staining, prosthesis survival and success, implant survival and success.

DETAILED DESCRIPTION:
The objectives of this randomized clinical trial are to 1) compare clinical performance of the two different treatment concepts during the follow up period of up to 3 years concerning prosthesis survival and success, 2) to assess the implants survival and success rates after 3 years, 3) to assess the accuracy of two surgical guides for full-arch implant surgery, 4) to assess the anticipated and actual pain following implant surgery, and 5) to assess patient satisfaction and quality of life will be assessed.

The study will be conducted according to the guidelines of the CONSORT statement for reporting randomized clinical. The study will be conducted at the College of Dental Medicine, University of Sharjah, United Arab Emirates.

Population and sample Study patients will be recruited from an existing pool of edentate adults referred for treatment to the College of Dental Medicine, University of Sharjah, United Arab Emirates. The patients will not be charged any treatment costs as part of this study. The target population will comprise patients requiring treatment for edentulous arches. Eligible patients for the implant phase of the study will be evaluated through a clinical assessment, panoramic radiograph, and cone-beam computed tomography (CBCT) exam. All study patients will be provided with a patient information sheet and provided written consent to take part in the study.

Conventional upper and lower denture constructions In the first phase of treatment, new maxillary and mandibular complete dentures with acceptable function and esthetics will be made and deliver to the patients. The conventional maxillary and mandibular complete denture constructions will follow the established methods which are primary impression with compound impression material, secondary impression with zinc oxide eugenol, jaw relation, try-in, issue and recall. The satisfactory mandibular complete denture will be converted into provisional all-on-4 mandibular prostheses immediately after implants placement.

Implant treatment planning The implant surgery planning will be performed using CBCT images of the anterior mandible obtained with a limited Field of View and standard protocols for minimizing radiation exposure. Implant placement planning and construction of surgical guides will be accomplished using available software and 3D printing machine. Implant placement will be fully guided surgery. The accuracy of two surgical guides will be assessed (milled and 3D-printed) by obtaining another CBCT after 3 months. The pre- and post-treatment scans will be superimposed and evaluated using Geomagic Control software.

Implant surgeries All implant surgeries will be performed by one surgeon. Surgeries will be carried out under local anesthesia. Four axial and tilted implants (All-on-4) will be placed in association with the treatment protocol. Four dental implants with a platform-switching design (Replace Conical Connection; Nobel Biocare, Zurich, Switzerland) will be placed with computer-guided technology (Nobel Guide; Nobel Biocare, Zurich, Switzerland) in the mandible at the lateral incisor and distal to first premolar sites. Primary stability of more than 35 Ncm will be achieved for all implants.

Pain Evaluation Anticipated pain will be recorded before surgery using visual analog scale (VAS) and actual pain levels will be recorded at day 1, 2 and 4 and at week 1, 2 and 3 after surgery using VAS.

Prostheses constructions Provisional prostheses Following implant placement, straight and 30-degree angled multiunit abutments will be torqued to the implants. Temporary abutments will be connected to the multiunit abutments, and the mandibular denture will be hollowed out to accommodate the temporary abutments. Rubber dam will be used to isolate the underlying soft tissue, and the temporary abutments will be connected to the denture with acrylic resin and picked up with the conversion prosthesis technique. The provisional prosthesis will be torqued to the multiunit abutments at 15 Ncm, and the screw access holes will be filled with Teflon tape and composite resin.

Definitive prostheses (conventional) Conventional hybrid prostheses combining metal frameworks as substructure, acrylic teeth and acrylic soft tissue will be constructed after three months of implants placement according to published protocols. Shimstock foil (GMH; Hanel Medizinal, Nu€rtingen, Germany) will be used for minor occlusal assessments during delivery of the prostheses. The prostheses will be torqued to the multi-unit abutments at 15Ncm, and the screw access holes will be filled with Teflon tape and composite resin (Z250, 3M ESPE, Minneapolis/St. Paul, MN). Oral hygiene instructions will be given to the patients. The follow up will be a week, three months, six months, a year, and 18 months or as needed by the patients. All prosthodontics procedures will be performed by the same prosthodontist.

Definitive prostheses (PEEK) Like conventional hybrid prostheses, the PEEK frameworks hybrid prostheses will also be constructed three months after implants' placement. The prostheses frameworks will be fabricated from modified PEEK (BioHPP; bredent GmbH & Co KG). The definitive impression will be made with a custom tray (Fastray LC; Harry J. Bosworth Co), medium viscosity polyether impression material (Impregum Penta; 3M ESPE), and low shrinkage auto polymerizing acrylic resin (GC pattern resin; GC America Inc) to splint the impression copings for better accuracy. The definitive cast will be poured with Type IV dental stone (Prima-Rock; Whip Mix Corp), and an accuracy transfer index will be fabricated on this cast. This index will be transferred intraorally to verify implant position. The implant misfit will be accommodated by sectioning the index and reconnecting it using the same low-shrinkage resin. This corrected position will be transferred onto the definitive cast by removing the analog from the cast and re-attaching and repositioning it with the transfer index in place. Once the accuracy of the definitive casts has been verified, a facebow transfer and an interocclusal centric relation record will be made using a conventional occlusal wax rim. The casts will be mounted on the semi-adjustable articulator (Denar Mark II; Whip Mix Corp). The cast with the implant abutments in place will be scanned with a laboratory scanner (Dental Create; Smart Optics GmbH); the implant framework will be digitally designed using digital software (Exocad; Exocad America Inc); and a wax implant framework pattern will be fabricated using CAD-CAM technology (DMU 80P duoBLOCK; DMG MORI). The wax frameworks will be made to fit over the selected abutments, which will be incorporated into the framework by using a sculpting wax (Thowax; Yeti Dental) and then cast in 1 piece from modified PEEK, using the conventional lost wax technique, using a special investment (Brevest; bredent GmbH & Co KG) and vacuum press device (2 press; bredent GmbH & Co KG) designed for this material. The fit of the PEEK framework will be verified intraorally, as is the space for the acrylic teeth and pink PMMA. The prostheses will clinically be evaluated to ensure correct tooth position, midline, esthetics, and phonetics. The PEEK framework will then be used to fabricate hybrid prostheses like conventional one. The implant supported prostheses will be tightened to 30 Ncm according to the manufacturer's instructions. Specific oral hygiene instructions will be given to the patients. The follow up will be a week, three months, six months, a year, and 18 months or as needed by the patients. All prosthodontic procedures will be performed by the same prosthodontist.

ELIGIBILITY:
Inclusion Criteria:

* no contraindications for implant surgery (including uncontrolled systemic diseases)
* sufficient bone height in the inter-foraminal area for an implant length of at least 10 mm
* ridge width of 5.5 mm for implant insertion of at least 3.5 mm in diameter,

Exclusion Criteria:

* individuals who disagreed with being randomly allocated to the treatment study groups, those with signs of untreated temporomandibular disorders or uncontrolled systemic or oral conditions requiring additional treatment, participants unable to understand and answer the questionnaires used in the study, and unable to attend the scheduled post-treatment appointments for longitudinal data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of full-arch surgical guides | 6 months
  Two types of surgical guides will be assessed for the accuracy. CBCT scans before and after surgery will be imported into 3D inspection software (Geomagic, 3D Systems Inc., Rock Hill, SC) for merging and evaluation of 3D deviations. Following software best-fit alignment, the 3D comparison will be used to evaluate the 3D deviations between the scans limited to the implants. Root man square (RMS) deviations will be recorded.
Survival rate of implants | 3 years
  Implant survival will be assessed clinically and radiographically every year. The criteria for implant success according to Buser et al, were no radiolucent zone around the implant, confirmed individual implant stability, and no suppuration, pain or ongoing pathologic processes (Buser et al., 1997). All implants that failed to fulfill these criteria will be regarded as failures.
Success rates of the Prostheses | 3 years
  Successful prosthesis must be free from any of the following technical complications: screw loosening, screw fracture, veneer material fracture or chipping, bulk fracture. Kaplan-meier analysis will be used.
Pain level | 1 months
  Anticipated and actual pain will be assessed before and after surgery using the 10-cm visual analog scale (VAS) ranging from 0 "no pain" to 10 "worst pain ever." The scale has no other markings along the line. Patients will be asked to record their pain level before surgery and after surgery, 24 hours after surgery, at day 2, day 4 and at week 1, week 2, and week 3.

SECONDARY OUTCOMES:
Marginal bone loss | 3 years
  Bone loss around implants will be measured radiographically every year for up to 3 years. All measurements will be done by one examiner, and radiographs will be analyzed using specially designed computer software (DicomWorks, Biomedical Engineering, the Netherlands) to perform linear measurements. Ideally, should be no bone loss, the higher the number after measurement the higher bone lost (resorbed) around implants.
Plaque index | 3 years
  The presence of plaque will be recorded using a plaque indicator liquid (Mira-2 Ton Liquid; Hager & Werken). The number of plaque sites will be analyzed according to modified plaque Index. Mild represents only 30% with plaque, moderate when up to 60% and severe when more than 60%.
Pocket depth | 3 years
  Pocket depth around implants will be meaured at baseline and every year using dental probe with light force (0.25 N). Pocket depths around healthy implants should generally be less than 5 mm in depth. Pockets more than 5 mm are indicative of an inflammation.
Bleeding index | 3 years
  Bleeding around implants will be assessed at baseline and every year using dental probe with light force (0.25 N) at six-points according to modified bleeding Index. Score 1 (up to 2 sites), score 2 (2-4 sites), score 3 (all sites).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Aziz, PhD, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Individuals data will not be shared, data required normally for publication will be shared upon reasonable request.

REFERENCES:
- [Background] Malo P, de Araujo Nobre M, Rangert B. Short implants placed one-stage in maxillae and mandibles: a retrospective clinical study with 1 to 9 years of follow-up. Clin Implant Dent Relat Res. 2007 Mar;9(1):15-21. doi: 10.1111/j.1708-8208.2006.00027.x. PMID 17362493
- [Background] Patzelt SB, Bahat O, Reynolds MA, Strub JR. The all-on-four treatment concept: a systematic review. Clin Implant Dent Relat Res. 2014 Dec;16(6):836-55. doi: 10.1111/cid.12068. Epub 2013 Apr 5. PMID 23560986
- [Background] Sailer I, Philipp A, Zembic A, Pjetursson BE, Hammerle CH, Zwahlen M. A systematic review of the performance of ceramic and metal implant abutments supporting fixed implant reconstructions. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:4-31. doi: 10.1111/j.1600-0501.2009.01787.x. PMID 19663946
- [Background] Fabbri G, Sorrentino R, Brennan M, Cerutti A. A novel approach to implant screw-retained restorations: adhesive combination between zirconia frameworks and monolithic lithium disilicate. Int J Esthet Dent. 2014 Winter;9(4):490-505. PMID 25289384
- [Background] Rubo JH, Capello Souza EA. Finite-element analysis of stress on dental implant prosthesis. Clin Implant Dent Relat Res. 2010 Jun 1;12(2):105-13. doi: 10.1111/j.1708-8208.2008.00142.x. Epub 2009 Feb 13. PMID 19220846
- [Background] Ciftci Y, Canay S. The effect of veneering materials on stress distribution in implant-supported fixed prosthetic restorations. Int J Oral Maxillofac Implants. 2000 Jul-Aug;15(4):571-82. PMID 10960992
- [Background] Davis DM, Rimrott R, Zarb GA. Studies on frameworks for osseointegrated prostheses: Part 2. The effect of adding acrylic resin or porcelain to form the occlusal superstructure. Int J Oral Maxillofac Implants. 1988 Winter;3(4):275-80. No abstract available. PMID 3075967
- [Background] Gracis SE, Nicholls JI, Chalupnik JD, Yuodelis RA. Shock-absorbing behavior of five restorative materials used on implants. Int J Prosthodont. 1991 May-Jun;4(3):282-91. PMID 1810320
- [Background] Stijacic T, Chung KH, Flinn BD, Raigrodski AJ. Effect of Tooth-Colored Restorative Materials on Reliability of Heat-Pressed Lithium Disilicate. J Prosthodont. 2015 Aug;24(6):475-83. doi: 10.1111/jopr.12243. Epub 2014 Dec 17. PMID 25522165